CLINICAL TRIAL: NCT00510185
Title: Italian Elderly ACS Study
Brief Title: Early Aggressive Versus Initially Conservative Therapy in Elderly Patients With Non-ST-Elevation Acute Coronary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Niguarda Hospital (Other)
Collaborators: Italian Society of Cardiology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Italian Elderly ACS Study
Record Dates: First submitted 2007-07-31; First posted 2007-08-01 (Estimated); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Acute Coronary Syndrome
Keywords: coronary artery disease; coronary angioplasty; coronary artery bypass surgery; elderly
MeSH Terms: conditions — Acute Coronary Syndrome; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Coronary angiography within 72h and revascularization as clinical indicated
  Interventions: Other: systematic coronary intervention
- 2 (Sham Comparator): Initially conservative treatment with coronary angiography only for recurrent ischemia
  Interventions: Other: coronary intervention only for cases refractory to medical therapy

INTERVENTIONS:
Other: systematic coronary intervention — Coronary angiography within 72 hrs
  Arms: 1
Other: coronary intervention only for cases refractory to medical therapy — Initially conservative treatment with coronary angiography only for recurrent ischemia
  Arms: 2

SUMMARY:
A randomized study comparing an early aggressive with an initially conservative strategy in patients >74 y.o. with non-ST-elevation acute coronary syndrome.

This study had generated a secondary one:

"Causes of death in elderly patients with Non-ST-Elevation Acute Coronary Syndrome; predictors of in-hospital and follow-up death"

DETAILED DESCRIPTION:
Patients >74 y.o. with non-ST-elevation acute coronary syndrome will be randomised to an early aggressive (coronary angiography within 72 hours followed, when indicated, by revascularization) or an initially conservative strategy (medical therapy, and coronary angiography only for refractory ischemia).

As reported in Amendment 1, the trial was stopped in May 2010 after the enrolment of 313 patients, which was the minimum sample size calculated in order to achieve a 80% power of detecting a difference in the primary-endpoint rate from 40% in the conservative arm to 25% in the invasive arm, based upon the log-rank test for survival curves (1-beta 0.80; 2-tailed alpha 0.05)

ELIGIBILITY:
Inclusion Criteria:

* Over 74 years of age.
* Have had symptoms suggestive of acute myocardial ischemia at rest within 48 hours prior to randomization, and ischemic ECG changes or elevated levels of biochemical markers of myocardial damage.
* Provide written informed consent before randomization.

Exclusion Criteria:

* Secondary causes of acute myocardial ischemia.
* Ongoing myocardial ischemia despite maximally titrated anti-ischemic therapy (invasive strategy recommended).
* Ongoing signs of acute heart failure despite treatment (invasive strategy recommended).
* Percutaneous coronary intervention or bypass surgery within 30 days prior to randomization.
* A serum creatinine level greater than 2.5 mg/dL.
* Active internal bleeding, history of hemorrhagic diathesis or recent transfusion of red blood cells, whole blood or platelets.
* History of cerebrovascular accident within the previous month.
* Known current platelet count < 90,000 cells/mL.
* Gastrointestinal or genitourinary bleeding of clinical significance within 6 weeks prior to randomization.
* Concomitant severe obstructive lung disease, malignancy or neurologic deficit limiting follow-up or adherence to the study protocol.
* Participation in any phase of another clinical research study involving the evaluation of another investigational drug or device within 30 days prior to randomization.
* Inability to give at least verbal informed consent to the study.

Min Age: 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 313 (Actual)
Dates: Start 2007-10; Primary Completion 2010-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
The composite of all-cause mortality, myocardial (re)infarction, disabling stroke and re-hospitalization for cardiovascular causes or severe bleeding within 1 yr. | 1 year

SECONDARY OUTCOMES:
CV mortality at 1 yr; All-causes mortality, myocardial re/infarction 1 yr; Composite of death, myocardial re/infarction, disabling stroke, rehospitalization due to cardiovascular or clinically bleeding causes at 1 yr; Major bleeding, stroke at 1 yr | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Savonitto, MD, Principal Investigator — Azienda Ospedaliera Ospedale Niguarda Ca' Granda-Dept. of Cardiology "A. De Gasperis"; Stefano De Servi, MD, Principal Investigator — Dept. of Cardiology - Ospedale Civile di Legnano - Italy
Locations (1):
- Dept. of Cardiology "A. De Gasperis", Milan, Italy

REFERENCES:
- [Background] Savonitto S, De Servi S, Petronio AS, Bolognese L, Cavallini C, Greco C, Indolfi C, Visconti LO, Piscione F, Ambrosio G, Galvani M, Marzocchi A, Santilli I, Steffenino G, Maseri A. Early aggressive vs. initially conservative treatment in elderly patients with non-ST-elevation acute coronary syndrome: the Italian Elderly ACS study. J Cardiovasc Med (Hagerstown). 2008 Mar;9(3):217-26. doi: 10.2459/JCM.0b013e3282f7c8df. PMID 18301136
- [Derived] Toso A, Servi SD, Leoncini M, Morici N, Murena E, Antonicelli R, Cavallini C, Petronio AS, Steffenino G, Piscione F, Bellandi F, Savonitto S. Acute Kidney Injury in Elderly Patients With Non-ST Elevation Acute Coronary Syndrome: Insights From the Italian Elderly: ACS Study. Angiology. 2015 Oct;66(9):826-30. doi: 10.1177/0003319714567738. Epub 2015 Jan 15. PMID 25593211
- [Derived] Savonitto S, Morici N, Cavallini C, Antonicelli R, Petronio AS, Murena E, Olivari Z, Steffenino G, Bonechi F, Mafrici A, Toso A, Piscione F, Bolognese L, De Servi S. One-year mortality in elderly adults with non-ST-elevation acute coronary syndrome: effect of diabetic status and admission hyperglycemia. J Am Geriatr Soc. 2014 Jul;62(7):1297-303. doi: 10.1111/jgs.12900. Epub 2014 Jun 10. PMID 24917216
- [Derived] Savonitto S, Cavallini C, Petronio AS, Murena E, Antonicelli R, Sacco A, Steffenino G, Bonechi F, Mossuti E, Manari A, Tolaro S, Toso A, Daniotti A, Piscione F, Morici N, Cesana BM, Jori MC, De Servi S; Italian Elderly ACS Trial Investigators. Early aggressive versus initially conservative treatment in elderly patients with non-ST-segment elevation acute coronary syndrome: a randomized controlled trial. JACC Cardiovasc Interv. 2012 Sep;5(9):906-16. doi: 10.1016/j.jcin.2012.06.008. PMID 22995877